Study Title: Double-Blinded Randomized Prospective Study On the Effects of Vitamin C, Hydrocortisone and Thiamine in Severe Sepsis and Septic Shock Patients.

October 25<sup>th</sup> 2017

#### **AIM OF OUR STUDY:**

The goal is to determine the effects on clinical course and outcome of patients with severe sepsis and septic shock treated with vitamin C, hydrocortisone and thiamine.

#### **BACKGROUND:**

This study will be conducted in the intensive care unit of Department of Gastroenterology, UMC Ljubljana. All of the patients with severe sepsis and septic shock admitted to the ICU in the past 12 hours will be screened for possible inclusion in the study. The diagnosis of severe sepsis and septic shock will be based on the 1992 American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference definitions.

## **PLAN OF THE STUDY:**

After determining the eligibility for inclusion in our study, we will acquire the written consent from the patient or relatives. We will randomize the patient either in the treatment or placebo group. The randomization will be done before-hand with the online tool Research Randomizer (online: https://www.randomizer.org). After acquiring the randomized numbers, they will be placed in sealed envelopes. These envelopes will be available to the on-call doctor. The envelopes will then be sent to our outpatient clinic, where the studied substances will be mixed by a nurse, that will have no contact with the patients or the ICU staff. The substances will be marked with Vitamin C, Thiamine and Hydrocortisone, regardless if normal saline or the actual substances are inside the vials. Only this nurse will have the data regarding the contents of the vials.

Vitamin C: Vitamin C will be mixed as 1500 mg vitamin C in 50ml container, which will then be infused over 30 minutes to 1 hour. The bag will be labeled by the pharmacy as Vitamin C. The dosing schedule is 1500mg every 6 hours for 4 days or until discharge from the ICU.

Vitamin C placebo will consist of an identical container of 50cc normal saline (but with no vitamin C) and will be labelled vitamin C. Placebo will be infused over 30-60 minutes as per the infusion instructions of the active vitamin.

Hydrocortisone: Hydrocortisone will be mixed as 50 mg of Hydrocortisone in 50 ml of 0.9 % Nalco. Patients will be treated with hydrocortisone 50mg IV q 6 hourly for 4 days or until ICU discharge.

Hydrocortisone placebo will be provided in an identical 50 ml bag of 0.9 % NaCl. Off label treatment with hydrocortisone or another corticosteroid will not be allowed.

Thiamine: Intravenous thiamine will be given in a dose of 200mg q 12 hourly for 4 days or until ICU discharge. Placebo patients will receive a matching vial of Normal Saline.

Based on literature we expect that survival and clinical course in sepsis and septic shock is correlated with fluid resuscitation and vasopressor use. Because of this, all of the included patients will be monitored with invasive hemodynamic monitoring (in our ICU we will be using the Edwards EV 1000 monitors).

All of the patients will be treated the same as per internationally recognized guidelines for treatment of septic shock. While the use of corticosteroids in severe sepsis is off-label, the patients will be informed of possible side-effects. This fact will also be written in the consent.

Neither the patients or the relatives will receive no financial compensation for study inclusion. During the hospitalization, the patients will receive three different substances in dosages, that are non toxic. During the study we will conduct intermittent statistical analysis, and if we would discover increased mortality or severe side effects, the study will be terminated. The confidentiality of personal data will be protected accordingly with the rules and laws of patient's privacy. The identity of patients will not be disclosed. The data acquired during the study will be available to the study participant. The anticipated costs will be covered by the Department of Gastroenterology, UMC Ljubljana. No financial compensation will be given to researchers.

## **INCLUSION CRITERIA:**

- I. Diagnosis of severe sepsis or septic shock within 12 hours of admission in our ICU.
- II. Informed consent.

## **EXCLUSION CRITERIA:**

- I. Age < 18 years
- II. Pregnancy
- III. DNR/DNI with limitations of care
- IV. Patients with fatal underlying disease who are unlikely to survive to hospital discharge (e.g.: disseminated malignant disease)
- V. Patients primarily admitted for acute coronary syndromes, acute cerebrovascular incidents or active GI bleeds
- VI. Patients that need immediate surgical treatment
- VII. Patients with HIV and a CD4 < 50 mm2,
- VIII Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency.
- IX. Patients with severe sepsis/septic shock transferred from another hospital
- X. Patients with features of sepsis/septic shock > 24 hours
- XI. Patients who require treatment with corticosteroids for an indication other than sepsis (chronic corticosteroid use, known Addison's Disease, Ulcerative colitis, Crohn's disease...)

# During the study we will be acquiring the following data from patients:

- 1. Age,
- 2. Sex,
- 3. Body weight,
- 4. Admitting diagnosis and source of infection,
- 5. Isolated pathogens,
- 6. Comorbidities,
- 7. The need for mechanical ventilation,
- 8. The use of vasopressors (all doses will be converted to Norepinephrine equivalents),
- 9. The duration of vasoactive therapy,
- 10. Daily urine output,
- 11. Fluid balance after 24 and 72 hours,
- 12. The presence of acute kidney failure
- 13. Duration of ICU stay and hospital stay,
- 14. Survival in ICU, hospital, after 28 and 60 days
- 15. Routine blood test for the first 4 days,
  - a. creatinine
  - b. WBC
  - c. Platelets
  - d. Bilirubin
  - e. PaO<sub>2</sub>/FiO<sub>2</sub> ration
  - e. procalcitonin (PCT) and procalcitonin clearens
  - f. lactate
  - g. blood samples will be stored for possible additional analysis

The patients' admission APACHE II and APACHE IV scores will be recorded. The APACHE IV score allows calculation of the predicted hospital mortality and predicted ICU length of stay (LOS). The daily SOFA (Sepsis-related Organ Failure Assessment) score will be recorded for the first 4 treatment days.

## STUDY END-POINTS:

# PRIMARY END-POINT

i. Hospital Mortality

## **SECONDARY END-POINTS**

- i. 60-day mortality
- ii. 28-day mortality
- iii. Time to vasopressor independence. Defined as the time from starting the active treatment/placebo to discontinuation of all pressors
- iv. PCT clearance (PCT-c) calculated using the following formula: initial PCT minus PCT at 96 hours, divided by the initial PCT multiplied by 100.
- v. Delta SOFA score, defined as the initial SOFA score minus the day 4 SOFA score vi. ICU mortality
- vii. ICU length of stay (LOS) and ICU free days. ICU free days is calculated as the number of days alive and out of the ICU to day 28
- viii. Hospital LOS

# **DATA ANALYSIS**

Summary statistics will be used to describe the clinical data and presented as mean ± SD, median with interquartile range (IQR) or percentages as appropriate. Chi squared analysis with Fisher's exact test (when appropriate) and Student's t test (Mann Whiney U test for non-normal distributions) were used to compare data between the active treatment group and the placebo group with statistical significance declared for probability values of 0.05 or less.

## **EXPECTED RESULTS:**

We expect a faster recovery, shorter hospitalization, shorter use of vasoactive drugs and better survival in treatment group vs. control group.

Sebastian Stefanovic, MD Department of Gastroenterology, UMC Ljubljana

#### References

- 1. Adhikari NK, Fowler RA, Bhagwanjee S et al. Critical care and the global burden of critical illness in adults. Lancet 2010; 376:1339-46.
- 2. Kaukonen KM, Bailey M, Suzuki S et al. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA 2014; 311:1308-16.
- 3. Gaieski DF, Edwards JM, Kallan MJ et al. Benchmarking the incidence and mortality of severe sepsis in the United States. Crit Care Med 2013; 41:1167-74.
- 4. Silva E, de Almeida Pedro M, Beltrami Sogayar AC et al. Brazilian Sepsis Epidemiological Study (BASES study). Crit Care 2004; 8:R251-R260.
- 5. Sales JA, David CM, Hatum R et al. Sepse Brasil: Estudo Epidemiologico da Sepse em Unidades de Terapia Intensiva Brasileiras. An epidemiological study of sepsis in Intensive Care Units. Sepsis Brazil Study. Rev Bras Ter Int 2006; 18:9-17.
- 6. The 10 leading causes of death by country income group 2012. WHO factsheets. <a href="http://www.who.int/mediacentre/factsheets/fs310/en/index1.html">http://www.who.int/mediacentre/factsheets/fs310/en/index1.html</a> . 2015. World Health Organization. 5-24-2016.
- 7. Wang HE, Szychowski JM, Griffin R et al. Long term mortality after sepsis. Chest 2013.
- 8. Artenstein AW, Higgins TL, Opal SM. Sepsis and scientific revolutions. Crit Care Med 2013; 41:2770-2772.
- 9. Fisher BJ, Seropian IM, Masanori Y et al. Ascorbic acid attenuates lipopolysaccharide-induced acute lung injury. Crit Care Med 2011; 39:1454-60.
- 10. Fisher BJ, Kraskauskas D, Martin EJ et al. Attenuation of sepsis-induced organ injury in mice by vitamin C. JPEN 2014; 38:825-39.
- 11. Han M, Pendem S, Teh SL et al. Ascorbate protects endothelial barrier function during septic insult: Role of protein phosphatase type 2A. Free Radic Biol Med 2010; 48:128.
- 12. Kim SR. Ascorbic acid reduces HMGB1 secretion in lipopolysaccharideactivated RAW 264.7 cells and improves survival rate in septic mice by activation of Nrf2/HO-1 signals. Biochemical Pharmacology 2015; 95:279-89.
- 13. Bornstein SR, Yoshida-Hiroi M, Sotiriou S et al. Impaired adrenal catecholamine system function in mice with deficiency of the ascorbic acid transporter (SVCT2). FASEB Journal 2003; 17:1928-30.

- 14. Wilson JX. Mechanism of action of vitamin C in sepsis: ascorbate modulates redox signaling in endothelium. Biofactors 2009; 35:5-13.
- 15. Wilson JX. Evaluation of vitamin C for adjuvant sepsis therapy. Antioxidants & Redox Signaling 2013; 19:2129-40.
- 16. Marik PE. Critical illness related corticoseroid insufficiency. Chest 2009; 135:181-93.
- 17. Annane D, Bellisant E, Bollaert PE et al. Corticosteroids for treating sepsis (Review). Cochrane Database of Syst Rev 2015.
- 18. Minneci PC, Deans KJ, Eichacker PQ et al. The effects of steroids during sepsis depend on dose and severity of illness: an updated meta-analysis. Clin Microbiol Infect 2009; 15:308-18.
- 19. Volbeda M, Wetterslev J, Gluud C et al. Glucocorticosteroids for sepsis: systematic review with meta-analysis and trial sequential analysis. Intensive Care Med 2015; 41:1220-1234.
- 20. Kalil AC, Sun J. Low-dose steroids for septic shock and severe sepsis; the use of Bayesian statistics to resolve clinical trial controversies. Intensive Care Med 2011; 37:420-429.
- 21. Sprung CL, Annane D, Keh D et al. Hydrocortisone therapy for patients with septic shock. N Engl J Med 2008; 358:111-24.
- 22. Nathens AB, Neff MJ, Jurkovich GJ et al. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg 2002; 236:814-22.
- 23. Fowler AA, Syed AA, Knowlson S et al. Phase 1 safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med 2014; 12:32.
- 24. Zabet MH, Mohammadi M, Ramezani M et al. Effect of high-dose ascorbic acid on vasopressor requirement in septic shock. J Res Pharm Pract 2016; 5:94-100.
- 25. Tanaka H, Matsuda T, Miyagantani Y et al. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg 2000; 135:326-31.
- 26. Ma Y, Chapman K, Levine M et al. High-dose parenteral ascorbate enhanced chemosensitivity of ovarian cancer and reduced toxicity of chemotherapy. Science Translational Medicine 2014; 6:222ra18.
- 27. Padayatty SJ, Rordan HH, Hewitt SM et al. Intravenously administered vitamin C as cancer therapy: three cases. CMAJ 2006; 174:937-42.
- 28. Hoffer LJ, Robitaille L, Zakarian R et al. High-dose intravenous vitamin C combined with cytotoxic chemotherapy in patients with advanced cancer: a phase I-II clinical trial. PloS ONE 2015; 10:e0120228.

- 29. Hoffer LJ, Levine M, Assouline S et al. Phase I clinical trial of i.v. ascorbic acid in advanced malignancy. Annals of Oncology 2008; 19:1969-74.
- 30. Stephenson CM, Levin RD, Spector T et al. Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetics of high-dose intravenous ascorbic acid in patients with advanced cancer. Cancer Chemotherapy & Pharmacology 2013; 72:139-46.
- 31. Monti DA, Mitchell E, Bazzan AJ et al. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PloS ONE 2012; 7:e29794.
- 32. Welsh JL, Wagner BA, van't Erve TJ et al. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol 2013; 71:765-75.
- 33. Ohno S, Ohno Y, Suzuki N et al. High-dose vitamin C (ascorbic acid) therapy in the treatment of patients with advanced cancer. Anticancer Research 2009; 29:809-15.
- 34. de Grooth HJ, Choo WP, Spoelstra-de Man AM et al. Pharmacokinetics of four high-dose regimens of intravenous Vitamin C in critically ill patients [Abstract]. Intensive Care Med 2016.
- 35. Padayatty SJ, Sun H, Wang Y et al. Vitamin C pharmacokinetics: implications for oral and intravenous use. Ann Intern Med 2004; 140:533-37.
- 36. Long CL, Maull KL, Krishman RS et al. Ascorbic acid dynamics in the seriously ill and injured. J Surg Res 2003; 109:144-48.
- 37. Ascorbic Acid Injection. <a href="http://www.drugs.com/pro/ascorbic-acid-injection.html">http://www.drugs.com/pro/ascorbic-acid-injection.html</a>
  . 2015. The Torrance Company. 6-12-2016.
- 38. Campbell GD, Steinberg MH, Bower JD. Ascorbic acid-induced hemolysis in G-6-PD deficiency [letter]. Ann Intern Med 1975; 82:810.
- 39. Rees DC, Kelsey H, Richards JD. Acute haemolysis induced by high dose ascorbic acid in glucose-6-phosphate dehydrogenase deficiency. BMJ 1993; 306:841-42.
- 40. Drouin G, Godin JR, Page B. The genetics of Vitamin C loss in vertebrates. Current Genomics 2011; 12:371-78.
- 41. Patak P. Vitamin C is an important cofactor for both adrenal cortex and adrenal medulla. Endocrine Research 2004; 30:871-75.
- 42. Das DD. Effect of vitamin C on adrenal suppression by etomidate induction in patients undergoing cardiac surgery: A randomized controlled trial. Ann Cardiac Anaesth 2016; 19:410.

- 43. Nooraei N, Fathi M, Edalat L et al. Effect of Vitamin C on serum cortisol after etomidate induction of anesthesia. J Cell Mol Anesth 2016; 1:28-33.
- 44. Massey LK. Ascorbate increases human oxaluria and kidney stone risk. Journal of Nutrition 2005; 135:1673-77.
- 45. Wandzilak TR. Effect of high dose vitamin C on urinary oxalate levels. Journal of Urology 1994; 151:834-37.
- 46. Hoppe B, Beck BB, Milliner D. The primary hyperoxalurias. Kidney Int 2009; 75:1264-71.
- 47. Sidhu H, Gupta R, Thind SK et al. Oxalate metabolism in thiamine-deficient rats. Ann Nutr Metab 1987; 31:354-61.
- 48. Ortiz-Alvarado O, Muyaoka R, Kriedberg C et al. Pyridoxine and dietary counseling for the management of idiopathic hyperoxaluria in stone-forming patients. Urology 2011; 77:1054-58.
- 49. Donnino MW, Andersen LW, Chase M et al. Randomized, double-blind, placebo-controlled trial of thiamine as a metabolic resuscitator in septic shock: A pilot study. Crit Care Med 2016; 44:360-367.
- 50. Moskowitz A, Anderson LW, Cocchi MN et al. Thiamine as a renal protective agent in septic shock: A secondary analysis of a randomized, double-blind, placebo-controlled trial. Ann Am Thorac Soc 2017;http://dx.doi.org/10.1513/AnnalsATS.201608-656BC.
- 51. Aird WC. The role of the endothelium in severe sepsis and multiple organ dysfunction syndrome. Blood 2003; 101:3765-77.
- 52. Marik PE, Pastores SM, Annane D et al. Recommendations for the diagnosis and management of corticosteroid insufficiency in critically ill adult patients: Consensus statements from an international task force by the American College of Critical Care Medicine. Crit Care Med 2008; 36:1937-49.
- 53. Okamoto K, Tanaka H, Makino Y et al. Restoration of the glucocorticoid receptor function by the phosphodiester compound of vitamins C and E, EPC-K1 (L-ascorbic acid 2-[3,4-dihydro-2,5,7,8-tetramethyl-2-(4,8,12-trimethyltridecyl)-2H-1-benzopyran-6-yl hydrogen phosphate] potassium salt), via a redox-dependent mechanism. Biochem Pharmacol 1998; 56:79-86.
- 54. Fujita I, Hirano J, Itoh N et al. Dexamethasone induces sodium-dependant vitamin C transporter in a mouse osteoblastic cell line MC3T3-E1. Br J Nutr 2001; 86:145-49.
- 55. Barabutis N, Khangoora V, Marik PE et al. Hydrocortisone and Ascorbic Acid synergistically protect against LPS-induced pulmonary endothelial barrier dysfunction. Chest 2017; Submitted.
- 56. Marik PE, Khangoora V, Rivera R et al. Hydrocortisone, Vitamin C and Thiamine for the treatment of severe sepsis and septic shock: A retrospective

- before-after study. Chest 2017; ePub:http://dx.doi.org/10.1016/j.chest.2016.11.036.
- 57. Marik PE. The physiology of volume resuscitation. Curr Anesthesiol Rep 2014; 4:353-59.
- 58. Marik PE. latrogenic salt water drowning and the hazards of a high central venous pressure. Ann Intensive Care 2014; 4:21.
- 59. Marik P, Bellomo R. A rational apprach to fluid therapy in sepsis. Br J Anaesth 2016; 116:339-49.
- 60. Marik PE. Fluid responsiveness and the six guiding principles of fluid resuscitation. Crit Care Med 2016; 44:1920-1922.
- 61. Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care 2016; 6:111.
- 62. Marik PE, Linde-Zwirble WT, Bittner EA et al. Fluid administration in severe sepsis and septic shock, patterns and outcomes. An analysis of a large national database. Intensive Care Med 2017; 43:625-32.
- 63. Society of Critical Care Medicine Consensus Conference Committee.

  American College of Chest Physicians/Society of Critical Care Medicine
  Consensus Conference: Definitions for sepsis and organ failure and
  guidelines for the use of innovative therapies in sepsis. Crit Care Med 1992;
  20:864-74.
- 64. Yealy DM, Kellum JA, Huang DT et al. A Randomized trial of protocol-based care for early septic shock. N Engl J Med 2014; 370:1683-93.
- 65. Mouncey PR, Osborn TM, Power S et al. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med 2015; 372:1301-11.
- 66. Peake SL, Delasney A, Bailey M et al. Goal-directed resuscitation for patients with Early Septic Shock. N Engl J Med 2014; 371:1496-506.
- 67. de Azevedo JR, Torres OJ, Beraldi RA et al. Prognostic evaluation of severe sepsis and septic shock: procalcitonin clearance vs DELTA Sequential Organ Failure Assessment. J Crit Care 2015; 30:219-12.
- 68. Ruiz-Rodriguez JC, Caballero J, Ruiz-Sanmartin A et al. Usefulness of procalcitonin clearance as a prognostic biomarker in septic shock. A prospective pilot study. Medicina Intensiva 2012; 36:475-80.
- 69. Flannery AH, Adkins DA, Cook AM. Unpeeling the evidence for the Banana Bag: Evidence-based recommendations for the management of alcohol-associated vitamin and electrolyte deficiencies in the ICU. Crit Care Med 2016; 44:1545-52.
- 70. Mancl EE, Muzevich KM. Tolerability and safety of enteral nutrition in critically ill patients receiving intravenous vasopressor therapy. JPEN 2013; 37:641-51.

- 71. Russell JA, Walley KR, Singer J et al. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med 2008; 358:877-87.
- 72. Knaus WA, Draper EA, Wagner DP et al. APACHE II: A severity of disease classification system. Crit Care Med 1985; 13:818-28.
- 73. Zimmerman JE, Kramer AA, McNair DS et al. Acute Physiology and Chronic Health Evaluation (APACHE) IV: hospital mortality assessment for today's critically ill patients. Crit Care Med 2006; 34:1297-310.
- 74. Vincent JL, Moreno R, Takala J et al. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med 1996; 22:707-10.
- 75. Ferreira FL, Bota DP, Bross A et al. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA 2001; 286:1754-58.